CLINICAL TRIAL: NCT04175405
Title: Low-level Laser Therapy With a 635nm Diode Laser Affects Orthodontic Mini-implants Stability. A Randomized Clinical Split-Mouth Trial.
Brief Title: Low-level Laser Therapy With a 635nm Diode Laser on Orthodontic Mini-implants Stability.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Jacek Matys, Principal Investigator, Wroclaw Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WroclawMU2212
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Malocclusion, Angle Class II
Keywords: ATP, biostimulation, micro-screw, Periotest, semiconductor laser
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — Lasers

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right side of the maxilla (Experimental): The 635-nm laser parameters; dose: 10J per point (20J/cm2), time: 100 sec per point, 2 points (irradiation on a buccal, and a palatal side of the alveolus/implant), the total energy per session 20J.
  Interventions: Procedure: Irradiation of implants with 635nm laser
- Left side of the maxilla (No Intervention)

INTERVENTIONS:
Procedure: Irradiation of implants with 635nm laser — Irradiation of implants with 635nm laser with a dose of 10J
  Arms: Right side of the maxilla

SUMMARY:
The study aimed to clinically estimate an influence of a 635nm diode laser on the primary and secondary stability of orthodontic mini-implants placed in a maxilla, to assess mini-implants failure rate (mini-implant loss) and to evaluate a pain level after the treatment. The randomized clinical split-mouth trial included 15 subjects, 30 implants (Dual Top Anchor System, Seoul, Korea) with a diameter 1.4mm and length of 10mm. Mini-implants were placed in the area of the attached gingiva between the second premolar and first molar teeth 2 mm below the mucogingival junction of both sides of the maxilla in 20 patients (13 women and 7 men; age: 32.5 ± 6.1 years).

ELIGIBILITY:
Inclusion Criteria:

* patients with class II malocclusion defect requiring lateral maxillary teeth distillation based on the use of orthodontic mini-implant;
* the patients were treated first time using fixed orthodontic appliance;
* no systemic diseases;
* were not using anti-inflammatory drugs;

Exclusion Criteria:

* had used antibiotics in the previous 24 months;
* smokers;
* had history of radiotherapy,
* taking bisphosphonate medication

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2019-06-02 (Actual); Study Completion 2019-10-24 (Actual)

PRIMARY OUTCOMES:
stability of orthodontic mini-implants | 60 days
  The mini-implants stability was estimated employing a Periotest device (Medzintechnik Gulden e K, Modautal, Germany). The Periotest measurement system includes the sound formed from contact between an object and a metallic tapping bar in a handpiece, which is electromagnetically driven and electronically verified. The Periotest response detection is analyzed through a fast Fourier transform (FFT) algorithm. Simply put, the Periotest answer to tapping is estimated by an accelerometer and then analyzed. The signal generated by tapping is then transformed to a value called the Periotest value (PTV), which depends on the damping characteristics of the peri-implant tissue. [27] The Periotest Test values (PTVs) are based on a numerical scale ranging from -8 to +50, defined by mathematical computation. The lower Periotest values indicate higher implant stability and thereupon the higher absorption effect of the target objects.

SECONDARY OUTCOMES:
Pain level | 24 hours
  Immediately after the mini-implants placement, each patient received a questionnaire for individual pain assessment (the numeric rating scale, NRS-11, grade level 0-10). The maximum pain level was measured at both sides of the maxilla during the first day after the treatment. The NRS-11 scale consists of a conscious, subjective assessment of the pain experienced; therefore, it is used in the case of patients over ten years old. A rating of 0 signifies no pain, 1-3 represents mild pain, 4-6 moderate pain, and 7-10 severe pain.
mini-implants loss | 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Private Dental Healtcare, Wschowa, Poland

IPD SHARING:
Plan to Share IPD: No